CLINICAL TRIAL: NCT05414656
Title: Comparison of Saddle Contoured Metal Matrix and Pre-contoured Self-adhesive Matrix in Composite Resin Class II Restorations
Brief Title: A Clinical Trial of Composite Class II Restorations With Two Different Matrix Bands
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, nosheen sarwar, Principle Investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOD/ERB/2022/02
Record Dates: First submitted 2022-06-02; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Class II Caries in Posterior Teeth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A : Saddle contoured metal matrix (Experimental): The prepared teeth received the Saddle contoured metal matrix. The saddle clip of matrix connect the band and secured around prepared cavity wall. The anatomical wedge placed into the gingival embrasure to maintain the height of gingival floor and ensure the optimal adaptation of the matrix band in the cervical region.
  Interventions: Device: Saddle contoured metal matrix, Pre-contoured self-adhesive matrix
- Group B:pre-contoured self-adhesive matrix (Active Comparator): Teeth received the Pre-contoured self adhesive matrix with anatomical wedges. The adhesive end of band closed around the prepared cavity.
  Interventions: Device: Saddle contoured metal matrix, Pre-contoured self-adhesive matrix

INTERVENTIONS:
Device: Saddle contoured metal matrix, Pre-contoured self-adhesive matrix — Saddle contoured metal matrix placed with the small clipper. The -contoured self-adhesive matrix has self adhesive ability.

SUMMARY:
Various procedures and techniques have been devised in an attempt to generate tighter and more anatomic proximal contacts with class II composite restorations. The investigators study focuses on using Saddle contoured metal matrix and pre-contoured self-adhesive matrix .Moreover, the investigators have attempted to study proximal tightness and proximal contours of composite restoration as separate variables.

DETAILED DESCRIPTION:
A total of 60 posterior teeth with proximal cavity to be assigned on alternate basis in two equal groups. Group A teeth received the Saddle contoured metal matrix and group B pre-contoured self-adhesive matrix after cavity preparation.

All teeth to be restored with Nano hybrid composite restorative material. Outcome of proximal contours and contact tightness is determined by a blinded assessor just after the restoration.

ELIGIBILITY:
Inclusion Criteria:

* • Permanent fully erupted teeth with class II supra-gingival caries or the necessity of replacing class II restoration.

  * The patient who has adjacent teeth available for the contact with surrounding tooth structure.
  * Teeth with cavity isthmus less than one-third of inter-cuspal distance

Exclusion Criteria:

* • Partially erupted or deciduous teeth.

  * Teeth with orthodontic bands or brackets.
  * 3rd Molar and rotated teeth.
  * Teeth with dental caries extending up to pulp with periapical pathosis or periodontally weak teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
proximal contacts tightness | immediately after procedure
  The tightness of the proximal contact area resulting from Saddle contoured metal matrix and pre-contoured self-adhesive matrix . It was measured using a nine inch long nylon dental floss (Oral-B, USA).

SECONDARY OUTCOMES:
Proximal contours and overhangs | immediately after procedure
  To be examined clinically with an explorer and mouth mirror and then on the radiograph by the blinded co investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarwar N, Khokhar SA. Comparison of saddle contoured metal matrix and pre-contoured self-adhesive matrix in composite resin class II restorations; an in vivo study. J Pak Med Assoc. 2024 Feb;74(2):209-215. doi: 10.47391/JPMA.8627. PMID 38419215